

# Statistical Analysis Plan

| Sponsor: | Terumo BCT, Inc. |
|---|---|
| Protocol No: | CTS-5085 |
| Protocol Title: | An In Vivo 24-Hour Recovery Study of<br>Leukoreduced RBCs After Automated<br>Separation of Whole Blood by the Reveos<br>System and Storage for 42 Days |
| Document Date: | 28-Apr-2022 |
| Document Revision | 1.0 |

Doc. No.: TMP-BS-01 Rev No.: 4.0



Revision No. 1.0

Document Date: 28-Apr-2022


# **APPROVAL SIGNATURES**

# Prosoft Personnel

| Title | Printed Name | Signature | Date |
|---|---|---|---|
| Manager,<br>Biostatistics | Christopher Dzura | DocuSigned by: Christopher Dzura | 28-Apr-2022 |
| | | Signer Name: Christopher Dzura Signing Reason: I am the author of th Signing Time: 28-Apr-2022 3:23:18 | |

D5BE1ABB694B4DF79A8F141B118D3B03

# Terumo BCT, Inc. Personnel

| Title | Printed Name | Signature | Date |
|---|---|---|---|
| Clinical Trial<br>Manager | Phillip Lopez, BS | DocuSigned by: Plulip Lopus Signer Name: Philip Lopez | 28-Apr-2022 |
| Sr. Clinical Research<br>Lead | Anna Maria<br>Neitenbach, MD | Signing Time: 28-Apr-2022 1:26:13 Boss A40Bd St 546058A7642EEC33 | E7EB9 |
| Sr. Manager Global<br>Clinical Affairs | Jack Rhodes, BS | Signing Reason: I approve this docum<br>Signing Time: 28-Apr-2022 1:48:49 F<br>As647711299F14647B3925B23D899 | ent<br>м2№0-тАрг-2022 |
| Consultant<br>Statistician | William Coar, PhD | Signer Name: Jack Rhodes Signing Reason: I approve this docun Signing Time: 29-Apr-2022 2:16:40 I 3BC40A2306EC41428DB19E05983 | M MDT |


Doc No.: TMP-BS-01 Rev No.: 4.0



Revision No. 1.0

Document Date: 28-Apr-2022


# **DOCUMENT HISTORY**

| Rev No | Date | Description |
|--------|-------------|-------------------|
| 1.0 | 28-APR-2022 | Original document |

Doc No.: TMP-BS-01 Rev No.: 4.0



Revision No. 1.0

Document Date: 28-Apr-2022


# TABLE OF CONTENTS

| 8 |
|----------|
| 8 |
| 8 |
| 8 |
| 8 |
| 9 |
| ALUATION |
| 9 |
| 10 |
| 11 |
| 11 |
| 12 |
| 12 |
| 12 |
| 12 |
| 12 |
| 12 |
| 13 |


Doc No.: TMP-BS-01

Rev No.: 4.0



Revision No. 1.0

Document Date: 28-Apr-2022


| 3. D | ATA HANDLING | 13 |
|-------|---------------------------------------------|----|
| 3.1 | Baseline and Study Visits | 13 |
| 3.2 | Missing, Unused, and/or Spurious Data | 13 |
| 3.3 | Incomplete Adverse Event Dates and/or Times | 13 |
| 3.4 | Incomplete Medication Dates | 13 |
| 4. Cl | HANGES FROM THE PROTOCOL | 14 |
| 5. RI | EFERENCES | 16 |


Doc No.: TMP-BS-01 Rev No.: 4.0



Revision No. 1.0

Document Date: 28-Apr-2022


# List of Abbreviations

| AABB | American Association of Blood Banks |
|--------|----------------------------------------------|
| ADE | adverse device effect |
| AE | adverse event |
| CIP | Clinical Investigation Plan |
| CIR | Clinical Investigation Report |
| FDA | United States Food and Drug Administration |
| IFU | Instructions for Use |
| LR-RBC | Leukoreduced red blood cell |
| MedDRA | Medical Dictionary for Regulatory Activities |
| PEAE | procedure-emergent adverse event |
| RBC | red blood cell |
| SAP | Statistical Analysis Plan |
| SAS | Statistical Analysis Software |
| SD | standard deviation |
| SOP | standard operating procedure |
| UADE | unanticipated adverse device effect |
| WB | whole blood |
| WBC | white blood cell |
| WHO | World Health Organization |


Doc No.: TMP-BS-01 Rev No.: 4.0



Revision No. 1.0

Document Date: 28-Apr-2022


#### 1. INTRODUCTION

### 1.1 Study Background

Blood transfusions have been widely used in medical practice since the early 20<sup>th</sup> century and are the most common procedure during hospital stays in the United States.<sup>[1,2]</sup> Patients may receive a unit of whole blood (WB) or individual blood components to treat any particular condition. Whole blood consists of blood components with cellular elements, colloids, and crystalloids.

Having different relative densities, sedimentation rate, and size, blood components can be separated when centrifugal force is applied. This separation is controlled in part by the specific gravities of these components including, in increasing order, plasma, platelets, leukocytes, and RBCs.<sup>[3]</sup>

The Reveos® Automated Blood Processing System (Reveos System) can process up to four (4) WB units in one run. It combines balancing, centrifugation, component separation, and sealing into one platform. As an automated blood processor, the Reveos System is beneficial in reducing manual blood processing drawbacks including processing time, and variability in the procedures and end product leading to standardized blood component yield and quality.

The aim of this study is to evaluate the in-vivo 24-hour recovery of autologous RBCs produced with the Reveos System and stored for 42 days, in order to meet the FDA's criteria for manufactured RBCs.

# 1.2 Study Design

This is a prospective, open label multicenter study to evaluate whether the LR-RBC derived from WB processing with the Reveos System meet FDA criteria for in vivo 24-hour recovery endpoints. Up to 50 healthy adult volunteers will be enrolled to target 24 evaluable recovery endpoints. Volunteers will be enrolled at 2 centers, with approximately 12 at each center.

An evaluable recovery endpoint is defined as having been collected from an enrolled participant that exhibits normal health status and vital signs as determined by standard American Association of Blood Banks (AABB) blood donation criteria and has also given appropriate informed consent, met all eligibility criteria, did not meet any exclusion criteria described in section 2.3 throughout the duration of the study, and did not have a change in health status which would cause them to fail the inclusion/exclusion criteria at the time of infusion.


Doc No.: TMP-BS-01 Rev No.: 4.0



Revision No. 1.0

Document Date: 28-Apr-2022


## 1.3 Study Objective

The primary objective of this study is to evaluate whether the LR-RBC derived from WB processed with the Reveos System meet FDA criteria for in vivo 24-hour recovery.

#### 1.4 Outcome Measures

# 1.4.1 Primary Endpoint

The primary endpoint is the 24-hour in vivo RBC recovery. The FDA criteria requires LR-RBC mean 24-hour recovery  $\geq$ 75% with standard deviation (SD)  $\leq$  9% and a one-sided lower confidence limit for the population proportion of RBCs in vivo recovery of 70% with a "success" being LR-RBC recovery >75%. This allows for low recoveries (<75%) in 2/20 or 3/24 volunteers.

#### 2. STATISTICAL METHODOLOGY

### 2.1 General Principles

All analyses will be performed using SAS® software version 9.4. Concomitant medications used to treat AEs will be coded using World Health Organization (WHO) Drug Dictionary Enhanced September 1, 2021 or later. Medical history and AEs will be coded using Medical Dictionary for Regulatory Activities (MedDRA) version 24.1 or later.

Inferential statistical tests will be identified in the post-text tables as being either one or two sided, and the construct of the confidence limits will be defined (e.g. 90% or 95%). A one-sided confidence interval for the proportion of subjects classified as a treatment success will be determined using an exact 95% confidence limit. Asymptotic confidence limits will be presented based on the normal approximation to the binomial distribution for all other presentations.

Continuous parameters will be summarized by n, mean, median, standard deviation (SD), minimum, and maximum. Except for efficacy parameters, 2-sided confidence limits will also be provided for continuous variables. Categorical variables will be summarized by count and percent. The following general conventions will be applied to all data presentations and analyses.

- All mean and median values will be formatted to one more decimal place than the measured value. Standard deviation values will be formatted to two more decimal places than the measured value. Minimum and maximum values will be presented with the same number of decimal places as the measured value
- The number and percentage of responses will be presented in the form XX (XX.X %) where the percentage is in the parentheses


Doc No.: TMP-BS-01 Rev No.: 4.0



Revision No. 1.0

Document Date: 28-Apr-2022


• All summary tables will include the analysis population sample size (i.e., number of subjects enrolled in the study)

# 2.2 Sample Size Determination

Up to 50 volunteers will be enrolled to allow targeted twenty-four (24) evaluable recovery endpoints.

In order to reach the total target number of evaluable subjects, additional subjects will be enrolled to replace subjects for whom the primary endpoints are not evaluable (i.e., those subjects who are lost-to-follow-up or withdrawn; those subjects whose health status has changed prior to their reinfusion, thereby potentially affecting their safety after receiving a reinfusion or potentially confounding study results; or those subjects for whom recovery calculations cannot be made due to missing value). All subjects, regardless of the availability of their endpoint data, will be included in evaluations of In vitro data (where samples are available) and in evaluations of AEs.

Estimates were prepared based on FDA criteria outlined in Section 1.4.1 with 24 subjects, examining the one-sided lower 95% confidence limit relative to the a priori value of 70%. Results are presented in the table presented below. If the observed proportion of treatment successes is 21/24 (87.50%) or higher, the one-sided lower 95% binomial confidence interval will exceed 70% (lower confidence limit = 70.77%).

Table 1: Statistical Scenarios 1-5 Estimation of LR-RBC Evaluation Sample Size

| Scenario Number | 1 | 2 | 3 | 4 | 5 | 6 |
|---|---|---|---|---|---|---|
| Number of Treatment<br>Successes | 17/24 | 18/24 | 19/24 | 20/24 | 21/24 | 22/24 |
| Percentage of Treatment Success | 70.83 | 75.00 | 79.17 | 83.33 | 87.50 | 91.67 |
| One-Sided Lower 95%<br>Confidence Limit | 52.13 | 56.53 | 61.09 | 65.82 | 70.77 | 76.02 |


Doc No.: TMP-BS-01 Rev No.: 4.0



| Statistical | <b>Analysis</b> | Plan | Template |
|-------------|-----------------|------|----------|

Revision No. 1.0

Document Date: 28-Apr-2022


Based on the binomial distribution, 24 evaluable LR-RBC products allow for 0, 1, 2 or 3 failures to establish 95% confidence that at least 70% of the products were successes.

If there are more than 24 evaluable recovery endpoints, then the allowable failure rate will be reevaluated to meet the FDA primary endpoint described in section 1.4.1. The following table shows the one-sided lower exact 95% confidence limits for the maximum allowable failure rate for different numbers of evaluable subjects.

Table 2: One-Sided Lower Exact 95% Confidence Limits for the Maximum Allowable Failure Rate

| Number of<br>Evaluable | Number of<br>Treatment<br>Successes | Number of<br>Treatment<br>Failures | Percentage of Success | Lower<br>Confidence<br>Limit |
|---|---|---|---|---|
| 24 | 21 | 3 | 87.50 | 70.77 |
| 25 | 22 | 3 | 88.00 | 71.83 |
| 26 | 23 | 3 | 88.46 | 72.81 |
| 27 | 24 | 3 | 88.89 | 73.73 |
| 28 | 24 | 4 | 85.71 | 70.23 |
| 29 | 25 | 4 | 86.21 | 71.16 |
| 30 | 26 | 4 | 86.67 | 72.01 |

# 2.3 Study Populations

The Full Analysis Population will include all participants enrolled in the study and who met the eligibility criteria. Efforts will be made to obtain complete recovery data from all participants.

The Safety Analysis Population will include all participants enrolled in the study who met the eligibility criteria and were exposed to Reveos Blood Bag Set. The Safety Analysis Population will be utilized to assess safety of the device and procedure. It is possible for a volunteer to be included in the Safety Analysis Population more than once if they do not have an evaluable


Doc No.: TMP-BS-01 Rev No.: 4.0



Revision No. 1.0

Document Date: 28-Apr-2022


recovery endpoint. If this occurs, it will be noted in the relevant tables in the Clinical Investigation Report (CIR) though they will continue to be analyzed as separate participants.

The Evaluable Analysis Population will include participants who completed all study visits per protocol with a valid 24-hour recovery endpoint. The Evaluable Analysis Population will be used in the analysis of the primary endpoint. While the criteria allow for 20 or 24 participants, analysis will be based on all participants meeting the criteria of the Evaluable Analysis Population.

Data will be excluded from the Evaluable Analysis Population in the following situations:

- 1. Incomplete or incorrect procedure that affects the primary endpoint due to:
  - a. Equipment failure or malfunction (eg, filter plugs)
  - b. Unanticipated processing failure
  - c. Results of primary endpoint tests are not available
- 2. Protocol deviations that affect the primary endpoint due to:
  - a. Failure to follow collection procedures outlined in the device Operator's Manual, Instructions for Use (IFU) (Package Insert), Manual of Procedure(s), and site SOPs
- 3. Product non-reinfusable due to:
  - a. Product does not pass quality check for reinfusion (residual WBC, LR-RBC mass recovery, visual inspection, hemolysis, bacterial growth)
- 4. Participant issues
  - a. Participant lost to follow-up or withdrawn from study
  - b. Other participant issues (eg, inadequate access, reaction, needle abort)

# 2.4 Participant Accounting and Baseline Characteristics

# 2.4.1 Participant Disposition

Enrollment and level of participation in the study will be summarized using the Full Analysis Population. The number and percent of participants per population will be summarized for each analysis population. The number and percentage of participants will also be presented for those participants who were screen failures or otherwise discontinued the study early and the reason for discontinuation will be noted.

Participant disposition data will be provided in a listing, which will cover each participant's eligibility for study participation as well as inclusion in or exclusion from each of the analysis populations (including enrollment and completion of study procedures, and/or evaluability).


Doc No.: TMP-BS-01 Rev No.: 4.0



Revision No. 1.0

Document Date: 28-Apr-2022


# 2.4.2 Participant Characteristics

Demographic and baseline characteristics will be provided in the listings for the Full Analysis Population and will be summarized for the Full Analysis Population, Safety Analysis Population, and Evaluable Analysis Population. Vital signs will be summarized for the Safety Analysis Population and laboratory results will be summarized for the Evaluable Analysis Population.

## 2.4.3 Clinical Investigation Plan Deviations

A listing of CIP deviations will be provided by the Sponsor.

#### 2.4.4 Device Deficiencies

A listing of Device Deficiencies will be provided by the Sponsor.

#### 2.5 Analyses

### 2.5.1 Primary Endpoint Analysis

The analysis of the primary endpoint will be conducted using the Evaluable Analysis Population.

The primary endpoint of RBC recovery at 24 hours post-infusion will be used to assess each of the three criteria specified by FDA. To assess the criteria associated with the percent of samples with at least a 75% recovery, a success or failure for each observed value will be determined. RBC recovery of at least 75% will be deemed a success, and failure otherwise. A one-sided confidence interval for the proportion of successes will be determined using the Clopper-Pearson exact method for a 95% confidence interval. If the one-sided 95% lower confidence limit is greater than 70% the study will have met its primary endpoint. Summary statistics will be presented to assess the actual RBC recovery values to evaluate the remaining criteria specified by FDA.

Primary endpoint will be reported with single label 24-hour endpoint recovery method. Dual label 24-hour recovery endpoint will also be reported as an exploratory method.

# 2.5.2 Safety Analyses

All adverse events collected will be provided for the Full Analysis Population by MedDRA system organ class and preferred term. Adverse event summaries for the purposes of device safety assessments will be limited to procedure-emergent adverse events (PEAEs), defined as any AE that occurs upon or after the exposure to the Reveos Blood Bag Set. PEAE summaries will be provided for the Safety Analysis Population.


Doc No.: TMP-BS-01 Rev No.: 4.0



Revision No. 1.0

Document Date: 28-Apr-2022


Tables will describe the frequency and percentage of all PEAEs, serious PEAEs, adverse device effects (ADEs), and unanticipated ADEs (UADEs). Additional presentations will summarize PEAEs by maximum reported severity; maximum relatedness to device, procedure, and medical history (related, not related); and those leading to discontinuation/termination. Concomitant medications used to treat PEAEs will also be summarized.

#### 2.5.3 Interim Analyses

No interim analyses are planned.

#### 3. DATA HANDLING

### 3.1 Baseline and Study Visits

Baseline is defined as the last non-missing scheduled assessment prior to first exposure and all other visits and time points are as recorded in the electronic case report forms except for early termination visits. Study participation will consist of 4 visits: Visit 1 for screening, Visit 2 for the WB collection, Visit 3 for reinfusion, and Visit 4 for assessing 24-hour RBC recovery percentage.

# 3.2 Missing, Unused, and/or Spurious Data

No imputation for missing, unused, and/or spurious data will be performed.

# 3.3 Incomplete Adverse Event Dates and/or Times

If an AE has an incomplete start date and/or time, the AE will be assumed to be a PEAE unless the provided dates/times or partial dates/times, if any, are enough to conclude that the AE could not have started on or after the start of the procedure.

# 3.4 Incomplete Medication Dates

In accordance with the CIP, reporting of concomitant medications is limited to those used to treat AEs. If a reported medication used to treat an AE has an incomplete start or stop date, the medication will be assumed to have been taken upon or after procedure initiation (ie, concomitant medication used to treat a PEAE) unless no PEAE was reported for the subject or the provided dates or partial dates, if any, are enough to conclude that the medication could not have been taken upon or after procedure initiation.


Doc No.: TMP-BS-01 Rev No.: 4.0



Revision No. 1.0

Document Date: 28-Apr-2022 

# 4. CHANGES FROM THE PROTOCOL

| | Summary of Changes | |
|---|---|---|
| Rationale: | This revision history captures the updates from Version 3.0 / 01 March 2022 of the CIP to Version 1.0 / 28-APR-2022 of the SAP. | |
| | Significant changes include the following: | |
| | <ol> <li>Changes and clarification were made to the definitions of the analysis populations.</li> <li>The sample size discussion was updated to accommodate over enrollment.</li> <li>The methods discussed for generating confidence intervals is inconsistent in the CIP. A one-sided lower exact 95% confidence limit will be provided for the proportion of treatment successes. Confidence limits presented for continuous demographic and safety parameters will be based on the normal approximation.</li> <li>Dual label method endpoint for 24-hour recovery will also be analyzed which include mean, standard deviation, median, minimum, maximum, proportion of successes, one-side 95% lower confidence limit.</li> <li>Administrative changes, section numbering, typographical error corrections, and minor wording changes for clarity, to make consistent throughout the text, or to make tables consistent with text as a result of these changes have been made and will not be reflected in the table below. These changes did not result in changes to the conduct of the study, so no CIP Amendment was conducted.</li> </ol> | |
| Change | Language from the CIP Language from the SAP | |
| Modification | 19.3.1 Full Analysis Population | Section 2.3 Study Populations |
| | The Full Analysis Population will include all participants enrolled in the trial. | The Full Analysis Population will include all participants enrolled in the study and who met the eligibility criteria. Efforts will be made to obtain complete recovery data from all participants. |
| Modification | 19.3.2 Safety Analysis PopulationThe Safety Analysis Population will include all participants enrolled in the trial who are exposed to Reveos Blood Bag Set and experience adverse event that is related to the device or study procedure as determined per; accordingly, the safety analysis will be limited to PEAEs (defined in Section 16.5). The Safety Analysis Population will be | Section 2.3 Study Populations The Safety Analysis Population will include all participants enrolled in the study who met the eligibility criteria and were exposed to Reveos Blood Bag Set. The Safety Analysis Population will be utilized to assess safety of the device and procedure. It is possible for a volunteer to be included in the Safety Analysis Population more than once if they do not have an evaluable |


Doc No.: TMP-BS-01 Rev No.: 4.0



Revision No. 1.0


Document Date: 28-Apr-2022

| | utilized to assess safety of the device and procedure. | recovery endpoint. If this occurs, it will be noted in the relevant tables in the Clinical Investigation Report (CIR) though they will continue to be analyzed as separate participants. |
|---|---|---|
| Modification | 19.3.3 Evaluable Analysis Population The analysis of the primary endpoint in the evaluable population will be based on all recorded data. Subjects are considered evaluable for the primary endpoints if they have: • Met all of the inclusion and none of the exclusion criteria at enrollment, • Were not found, after being enrolled in good faith, to be in fact, non-compliant with one or more of the inclusion/exclusion criteria, • The subject has not had a change in health status which would cause them to fail the inclusion/exclusion criteria at the time of infusion of radiolabeled cells • Have not met any other protocol exclusion criteria as defined in Section 19.4. The Evaluable Analysis Population will be included in the analysis of the primary endpoint. Within the enrolled population, all attempts will be made to obtain complete recovery data from all subjects for the analysis of the primary endpoint. | Section 2.3 Study Populations The Evaluable Analysis Population will include all participants who completed all study visits per protocol with a valid 24-hour recovery endpoint. The Evaluable Analysis Population will be used in the analysis of the primary endpoint. While the criteria allow for 20 or 24 participants, analysis will be based on all participants meeting the criteria of the Evaluable Analysis Population. |
| Added | | Section 2.2 Sample Size Determination Based on the binomial distribution, 24 evaluable |
| | | LR-RBC products allow for 0, 1, 2 or 3 failures to establish 95% confidence that at least 70% of the products were successes. |
| | | If there are more than 24 evaluable recovery endpoints, then the allowable failure rate will be |


Doc No.: TMP-BS-01 Rev No.: 4.0



Revision No. 1.0

Document Date: 28-Apr-2022 

| | | shows the limits for different | d in sect<br>ne one-si<br>r the ma<br>t number | tion 1.4. ided low eximum rs of eva | .1. The foregraph of the second secon | following t 95% co le failure subjects. | - |
|---|---|---|---|---|---|---|---|
| Revised | Section 19 Statistical Plan Asymptotic confidence limits will be presented based on the normal approximation to the binomial distribution for the proportion of subjects classified as a treatment success. Exact confidence intervals will be used for all other presentations. | Section 2.1 General Principles A one-sided confidence interval for the proportion of subjects classified as a treatment success will be determined using an exact 95% confidence limit. Asymptotic confidence limits will be presented based on the normal approximation to the binomial distribution for a other presentations. Section 2.5.1 Primary Endpoint Analysis A one-sided confidence interval for the proportion of successes will be determined using the Clopper-Pearson exact method for a 95% confidence interval. | | et 95% e limits on for all | | | |
| Revised | Section 19.2.1 Primary Endpoint Additional exploratory analyses may be performed on estimates of RBC recovery using RBC mass derived from 99mTc radiolabeling. | Section 2.5.1 Primary Endpoint Analysis Primary endpoint will be reported with single label 24-hour endpoint recovery method. Dual label 24-hour recovery endpoint will also be reported as an exploratory method. | | | | | |

# 5. REFERENCES

<sup>1</sup> Yaddanapudi S, Yaddanapudi L. Indications for blood and blood product transfusion. Indian J Anaesth.

#### Confidential Document

Doc No.: TMP-BS-01 Rev No.: 4.0



Revision No. 1.0

Document Date: 28-Apr-2022


2014;58(5):538-542.

<sup>2</sup> Pfuntner A, Wier LM, Stocks C. Most frequent procedures performed in U.S. hospitals, 2010. HCUP statistical


Doc No.: TMP-BS-01 Rev No.: 4.0

<sup>&</sup>lt;sup>3</sup>Basu D, Kulkarni R. Overview of blood components and their preparation. Indian J Anaesth. 2014;58(5):529-537.

# **DocuSign**

#### **Certificate Of Completion**

Envelope Id: D0862A39F2484B5D88B5A5248064F831

Subject: Please DocuSign: CTS-5085\_SAP v1.0 28APR2022.pdf

Source Envelope:

Document Pages: 17 Signatures: 4
Certificate Pages: 6 Initials: 0

AutoNav: Enabled

**Envelopeld Stamping: Disabled** 

Time Zone: (UTC-05:00) Eastern Time (US & Canada)

Status: Sent

Envelope Originator: Christopher Dzura 996 Old Eagle School Rd

**Suite 1106** 

Wayne, PA 19087

Location: DocuSign

c.dzura@prosoftclinical.com IP Address: 71.224.170.54

Sent: 4/28/2022 3:22:22 PM

Viewed: 4/28/2022 3:23:01 PM

Signed: 4/28/2022 3:23:28 PM

Sent: 4/28/2022 3:23:30 PM

Viewed: 4/28/2022 3:25:43 PM

Signed: 4/28/2022 3:26:17 PM

#### **Record Tracking**

Status: Original

4/28/2022 3:03:42 PM

Holder: Christopher Dzura

c.dzura@prosoftclinical.com

# Timestamp

Signer Events
Christopher Dzura

c.dzura@prosoftclinical.com

Manager Biostatistics

Prosoft Clinical

Security Level: Email, Account Authentication

(Required)

Christopher Dzura

Signature Adoption: Pre-selected Style

Signed by link sent to c.dzura@prosoftclinical.com

Signature ID:

Signature

D5BE1ABB-694B-4DF7-9A8F-141B118D3B03

Using IP Address: 71.224.170.54

With Signing Authentication via DocuSign password

With Signing Reasons (on each tab):

I am the author of this document

#### **Electronic Record and Signature Disclosure:**

Accepted: 5/26/2020 9:06:13 AM

ID: 3fb957da-aaae-4b12-b819-ea918e01af3b

Philip Lopez

phillip.lopez@terumobct.com

Security Level: Email, Account Authentication

(Required)

DocuSigned by:

Philip lopes

Signer Name: Philip Lopez Signing Reason: I approve this document Signing Time: 28-Apr-2022 | 1:26:13 PM MDT

-B5B8A40B03E546058A7642EEC33E7EB9

Signature Adoption: Pre-selected Style

Signed by link sent to phillip.lopez@terumobct.com

Signature ID:

B5B8A40B-03E5-4605-8A76-42EEC33E7EB9

Using IP Address: 208.51.143.189

With Signing Authentication via DocuSign password

With Signing Reasons (on each tab):

I approve this document

#### **Electronic Record and Signature Disclosure:**

Accepted: 4/28/2022 3:25:43 PM

ID: 8698f9ea-2414-4fa4-9e8f-4faf1dc6a947

**Signer Events** 

Anna Maria Neitenbach annamaria.neitenbach@terumobct.com

Security Level: Email, Account Authentication (Required)

Signature

–DocuSigned by: Unna Maria Mitenbadu

U

Signer Name: Anna Maria Neitenbach Signing Reason: I approve this document Signing Time: 28-Apr-2022 | 1:48:49 PM MDT

-A36477FE99F14647B3925B23D899C445

Signature Adoption: Pre-selected Style

Signed by link sent to

annamaria.neitenbach@terumobct.com

Signature ID:

A36477FE-99F1-4647-B392-5B23D899C445

Using IP Address: 208.51.143.189

With Signing Authentication via DocuSign password

With Signing Reasons (on each tab):

I approve this document

**Electronic Record and Signature Disclosure:** 

Accepted: 4/28/2022 3:48:07 PM

ID: 395b416a-818f-480d-816e-4d32e7b924b0

Jack Rhodes

jack.rhodes@terumobct.com

Security Level: Email, Account Authentication

(Required)

Jack Phodes

Sent: 4/28/2022 3:49:04 PM Viewed: 4/29/2022 4:16:23 PM Signed: 4/29/2022 4:16:44 PM

**Timestamp** 

Sent: 4/28/2022 3:26:20 PM

Viewed: 4/28/2022 3:48:07 PM

Signed: 4/28/2022 3:49:01 PM

Signature Adoption: Pre-selected Style

Signed by link sent to jack.rhodes@terumobct.com

Signature ID:

3BC40A23-06EC-4142-8DB1-9E059837B6D9

Using IP Address: 208.51.143.189

With Signing Authentication via DocuSign password

With Signing Reasons (on each tab):

I approve this document

**Electronic Record and Signature Disclosure:** 

Accepted: 4/29/2022 4:16:23 PM ID: dcff30d1-01af-4ed1-883e-41d932246538

William Coar

william.coar@cytel.com

Security Level: Email, Account Authentication

(Required)

**Electronic Record and Signature Disclosure:** 

Not Offered via DocuSign

Sent: 4/29/2022 4:16:47 PM

| In Person Signer Events | Signature | Timestamp |
|------------------------------|-----------|-----------|
| Editor Delivery Events | Status | Timestamp |
| Agent Delivery Events | Status | Timestamp |
| Intermediary Delivery Events | Status | Timestamp |
| Certified Delivery Events | Status | Timestamp |
| Carbon Copy Events | Status | Timestamp |
| Witness Events | Signature | Timestamp |

| Notary Events | Signature | Timestamp |
|---|---|---|
| Envelope Summary Events | Status | Timestamps |
| Envelope Sent | Hashed/Encrypted | 4/28/2022 3:22:22 PM |
| Payment Events | Status | Timestamps |
| Electronic Record and Signature Disclosure | | |

#### ELECTRONIC RECORD AND SIGNATURE DISCLOSURE

From time to time, Prosoft Clinical (we, us or Company) may be required by law to provide to you certain written notices or disclosures. Described below are the terms and conditions for providing to you such notices and disclosures electronically through the DocuSign system. Please read the information below carefully and thoroughly, and if you can access this information electronically to your satisfaction and agree to this Electronic Record and Signature Disclosure (ERSD), please confirm your agreement by selecting the check-box next to 'I agree to use electronic records and signatures' before clicking 'CONTINUE' within the DocuSign system.

#### Getting paper copies

At any time, you may request from us a paper copy of any record provided or made available electronically to you by us. You will have the ability to download and print documents we send to you through the DocuSign system during and immediately after the signing session and, if you elect to create a DocuSign account, you may access the documents for a limited period of time (usually 30 days) after such documents are first sent to you. After such time, if you wish for us to send you paper copies of any such documents from our office to you, you will be charged a \$0.00 per-page fee. You may request delivery of such paper copies from us by following the procedure described below.

#### Withdrawing your consent

If you decide to receive notices and disclosures from us electronically, you may at any time change your mind and tell us that thereafter you want to receive required notices and disclosures only in paper format. How you must inform us of your decision to receive future notices and disclosure in paper format and withdraw your consent to receive notices and disclosures electronically is described below.

#### Consequences of changing your mind

If you elect to receive required notices and disclosures only in paper format, it will slow the speed at which we can complete certain steps in transactions with you and delivering services to you because we will need first to send the required notices or disclosures to you in paper format, and then wait until we receive back from you your acknowledgment of your receipt of such paper notices or disclosures. Further, you will no longer be able to use the DocuSign system to receive required notices and consents electronically from us or to sign electronically documents from us

#### All notices and disclosures will be sent to you electronically

Unless you tell us otherwise in accordance with the procedures described herein, we will provide electronically to you through the DocuSign system all required notices, disclosures, authorizations, acknowledgements, and other documents that are required to be provided or made available to you during the course of our relationship with you. To reduce the chance of you inadvertently not receiving any notice or disclosure, we prefer to provide all of the required notices and disclosures to you by the same method and to the same address that you have given us. Thus, you can receive all the disclosures and notices electronically or in paper format through the paper mail delivery system. If you do not agree with this process, please let us know as described below. Please also see the paragraph immediately above that describes the consequences of your electing not to receive delivery of the notices and disclosures electronically from us.

#### **How to contact Prosoft Clinical:**

You may contact us to let us know of your changes as to how we may contact you electronically, to request paper copies of certain information from us, and to withdraw your prior consent to receive notices and disclosures electronically as follows:

To contact us by email send messages to: t.sammartino@prosoftclinical.com

#### To advise Prosoft Clinical of your new email address

To let us know of a change in your email address where we should send notices and disclosures electronically to you, you must send an email message to us at t.sammartino@prosoftclinical.com and in the body of such request you must state: your previous email address, your new email address. We do not require any other information from you to change your email address.

If you created a DocuSign account, you may update it with your new email address through your account preferences.

#### To request paper copies from Prosoft Clinical

To request delivery from us of paper copies of the notices and disclosures previously provided by us to you electronically, you must send us an email to t.sammartino@prosoftclinical.com and in the body of such request you must state your email address, full name, mailing address, and telephone number. We will bill you for any fees at that time, if any.

#### To withdraw your consent with Prosoft Clinical

To inform us that you no longer wish to receive future notices and disclosures in electronic format you may:

i. decline to sign a document from within your signing session, and on the subsequent page, select the check-box indicating you wish to withdraw your consent, or you may;

ii. send us an email to t.sammartino@prosoftclinical.com and in the body of such request you must state your email, full name, mailing address, and telephone number. We do not need any other information from you to withdraw consent. The consequences of your withdrawing consent for online documents will be that transactions may take a longer time to process.

#### Required hardware and software

The minimum system requirements for using the DocuSign system may change over time. The current system requirements are found here: <a href="https://support.docusign.com/guides/signer-guide-signing-system-requirements">https://support.docusign.com/guides/signer-guide-signing-system-requirements</a>.

#### Acknowledging your access and consent to receive and sign documents electronically

To confirm to us that you can access this information electronically, which will be similar to other electronic notices and disclosures that we will provide to you, please confirm that you have read this ERSD, and (i) that you are able to print on paper or electronically save this ERSD for your future reference and access; or (ii) that you are able to email this ERSD to an email address where you will be able to print on paper or save it for your future reference and access. Further, if you consent to receiving notices and disclosures exclusively in electronic format as described herein, then select the check-box next to 'I agree to use electronic records and signatures' before clicking 'CONTINUE' within the DocuSign system.

By selecting the check-box next to 'I agree to use electronic records and signatures', you confirm that:

- You can access and read this Electronic Record and Signature Disclosure; and
- You can print on paper this Electronic Record and Signature Disclosure, or save or send this Electronic Record and Disclosure to a location where you can print it, for future reference and access; and
- Until or unless you notify Prosoft Clinical as described above, you consent to receive
  exclusively through electronic means all notices, disclosures, authorizations,
  acknowledgements, and other documents that are required to be provided or made
  available to you by Prosoft Clinical during the course of your relationship with Prosoft
  Clinical.